CLINICAL TRIAL: NCT03785236
Title: Visualizing Beta Cells After Intrahepatic Islet of Langerhans Transplantation
Brief Title: Visualizing Beta Cells After Islet Transplantation
Acronym: GLP1-transpl
Status: Terminated | Type: Observational
Why Stopped: Suitable participants have complicated T1D, often with serious complications, participation is therefore challenging. Participants also fall within an unique group and few suitable individuals were available for inclusion.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL52630.091.15
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tx-group: T1D patients that received islet of Langerhans transplantation (Tx) at least 3 months earlier
  Interventions: Radiation: 68Ga-NODAGA-exendin PET/CT
- Control group: T1D patients that await islet of Langerhans transplantation
  Interventions: Radiation: 68Ga-NODAGA-exendin PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin PET/CT — 68Ga-NODAGA-exendin PET/CT

SUMMARY:
In patients with type 1 diabetes (T1D) that have undergone islet of Langerhans transplantation or are on the waiting list for transplantation, Ga-68-exendin PET imaging is performed to study the visualization of transplanted islet grafts in patients.

DETAILED DESCRIPTION:
Detecting damage to islets with a reliable imaging technique could be important for improving islet survival after transplantation. This could lead to better patient outcomes which would be of great interest for the treatment of type 1 diabetes. In order to assess the possibility of visualizing transplanted islet grafts with Ga-68-NODAGA-exendin-4 PET, a proof-of -concept study is performed in 10 patients with type 1 diabetes who have undergone intrahepatic islet transplantation with biochemically proven functional islet grafts and 5 patients with type 1 diabetes who are on the waiting list for islet transplantation. The investigators propose to determine the uptake of the radiolabeled tracer and compare it to functionality of the islet grafts. These highly relevant data will provide us with more information on the suitability of GLP-1 receptor imaging for monitoring of transplanted islet mass.

ELIGIBILITY:
Inclusion Criteria

Tx-group:

* >18 years old
* T1D patient undergone islet transplantation
* Clinically proven functional islet graft
* Signed informed consent

Control group:

* >18 years old
* T1D patients who are on the waiting list for islet transplantation
* Signed informed consent

Exclusion Criteria:

* Treatment with synthetic exendin or Dipeptidyl-Peptidase IV inhibitors within the last 3 months
* Breast feeding
* Pregnancy or the wish to become pregnant within 6 months
* Kidney disease
* Liver disease
* Age <18 years
* No signed informed consent

Exclusion criteria for MR:

* fragments, clips or devices in brain, eyes, spinal canal
* Implantable defibrillator or pacemaker (wires)
* Mandibular magnetic implants
* Neurostimulator, bladder stimulator, non-removable insulin pump
* Metal tissue-expander in chest
* Cochlear implant
* Ossicular replacement prosthesis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population consists of 10 individuals with type 1 diabetes patients who have undergone intrahepatic islet transplantation at least 3 months earlier at. Furthermore, 5 T1D patients without an islet transplant will be included as a control for uptake of the radiotracer in the liver. All participating individuals need to be 18 years or older. In total, 15 participants will be included.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Hepatic uptake of 68Ga-NODAGA-exendin-4 | 1 year
  Hepatic uptake of 68Ga-NODAGA-exendin-4 obtained by quantitative analysis

SECONDARY OUTCOMES:
Islet graft function | 1 year
  Correlation of tracer uptake and islet graft function

CONTACTS AND LOCATIONS:
Locations (2):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No